CLINICAL TRIAL: NCT06595537
Title: Gastric Ultrasound Feeding Tube Placement Confirmation Study
Acronym: GUT
Status: Recruiting | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, jelopezmatta, Medical Doctor, Leiden University Medical Center
Other Study IDs: NL77930.058.21
Record Dates: First submitted 2024-01-12; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Gastric Feeding Tubes; Ultrasound
Keywords: gastric ultrasound; Gastric feeding tube; Point of care ultrasound

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Ultrasound control of air insufflation in tracheobronchial suction catheter, oesofagus and stomach: Patients will receive a gastric feeding tube. At mid-esophagus level and at gastric level, placement of the gastric feeding tube will be controlled through doppler-ultrasound after air-insufflation. Ultrasound control after air insufflation will also take place after placing a suction catheter through the endotracheal tube in the trachea. Finally the gastric feeding tube placement will be confirmed with chest X-ray.
  Interventions: Device: Hand held ultrasound

INTERVENTIONS:
Device: Hand held ultrasound — Determination of gastric feeding tube position with the use of Lumify handheld ultrasound
  Other Names: Lumify handheld ultrasound

SUMMARY:
Objective

This study aims to assess the accuracy and reliability of ultrasound in determining the correct placement of gastric feeding tubes (GFTs) in intensive care patients.

Study Design

A diagnostic study will be conducted to evaluate the efficacy of ultrasound in determining GFT placement in all ICU patients who require GFT placement. Patients will undergo ultrasound by an ultrasonographer (USG) after receiving a new or replaced GFT. The USG will assess the presence or absence of a "mosaic sign" after insufflation of 20 mL of air through the GFT. The mosaic sign indicates proper GFT placement in the stomach.

Methods

All ultrasonographic measurements will be recorded and saved in a central picture archiving and communication system (PACS). The images will be labeled with the deepness of the GFT (20 cm, 50 cm, or tracheobronchial) and anonymized before being presented to an intensivist expert in USG for interpretation.

Hypothesis

A 20 mL air insufflation via a GFT at the esophageal level or via a suction catheter in the tracheobronchial system will not produce a "mosaic sign" on ultrasound. This sign will only be present if the GFT is properly positioned in the stomach.

DETAILED DESCRIPTION:
Objective: To evaluate the effectiveness of ultrasound Doppler in determining the correct placement of gastric feeding tubes (GFTs) in intensive care patients compared to the standard of care, chest X-ray (CXR).

Study Design: A diagnostic study involving ICU patients who require GFT placement or replacement.

Background: Misplacement of GFTs is a common complication in ICU settings, with significant potential consequences for patient safety. Ultrasound Doppler has emerged as a potential alternative to CXR for confirming GFT placement due to its portability, ease of use, and real-time assessment.

Methods:

Subject Selection: Subjects will be recruited from the ICU at the Leiden University Medical Center (LUMC) who meet the inclusion criteria: tracheally intubated, require GFT placement or replacement, and provide informed consent.

Ultrasound Procedure: At the esophageal and gastric levels, ultrasound will be performed using a Philips Lumify® S4-1 broad band sector array transducer. An antrum Doppler window will be set to visualize the "mosaic sign," a characteristic Doppler signal indicative of correct GFT placement.

Image Acquisition and Coding: During ultrasound, 20 ml of air will be injected through the GFT, and images will be captured. These images will be anonymized and labeled with the depth at which the insufflation occurred (20 cm or 50 cm) or the location of the insufflation (tracheal suction catheter).

Ultrasound Interpretation: An intensivist expert in ultrasound will blind to the original localization of the GFT analyze the anonymized images. The intensivist will classify each image as having a "mosaic sign present" or "mosaic sign absent."

Correlation with CXR: The ultrasound interpretation will be compared to the gold standard of CXR to determine the sensitivity and specificity of ultrasound Doppler.

Secondary Objectives:

* Investigate the correlation between false positive and false negative results and patient characteristics such as gender, BMI, positive end-expiratory pressure (PEEP), tidal volume, and presence of abdominal gas in CXR.
* Assess the safety of ultrasound Doppler in terms of adverse events (AEs) and serious adverse events (SAEs).

Sample Size: A sample size of 58 patients is expected to provide sufficient power to detect statistically significant differences in sensitivity and specificity between ultrasound Doppler and CXR.

Ethical Considerations:

Ethical Approval: The study protocol has been approved by the Leiden University Medical Center Ethical Review Board (LUMC-ERB).

Informed Consent: All participants will provide informed consent prior to undergoing ultrasound Doppler and CXR.

Safety Monitoring: Adverse events will be monitored and reported as per the regulations of the LUMC and the Medical Research Involving Human Subjects Act (WMO).

Administrative Aspects:

Data Collection and Storage: Patient and clinical data, including anonymized ultrasound images and CXRs, will be collected and stored using the Castor cloud-based clinical data management system.

Monitoring: The study will be monitored by internal monitors of the Leiden University Medical Center (LUMC).

Reporting: Annual progress reports will be submitted to the accredited METC, and the final study report will be submitted upon completion of the study.

Expected Findings:

Ultrasound Doppler is expected to demonstrate high sensitivity and specificity in determining the correct placement of GFTs in ICU patients compared to CXR.

Potential correlation between false positive and false negative results with certain patient characteristics, such as gender, BMI, and presence of abdominal gas in CXR, may be identified.

The safety profile of ultrasound Doppler is expected to be favorable with minimal AEs and no SAEs.

Conclusion: This study aims to evaluate the efficacy of ultrasound Doppler in determining the correct placement of GFTs in ICU patients. The findings of this study will contribute to the development of non-invasive methods for confirming GFT placement, potentially improving patient safety and reducing the need for CXRs.

ELIGIBILITY:
Inclusion Criteria:

* Being tracheally intubated

  * Have a gastric feeding tube which needs replacement for any particular reason e.g the GFT is not functioning, has been displaced, and the patient has no exclusion criteria ( zie 4.3).
  * Need a gastric feeding tube
  * Given informed consent directly

Exclusion Criteria:

* Does not need a gastric feeding tube and doesn't have one.
* Laparotomy wound interfering with abdominal ultrasound.
* Patient in prone position
* No informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of tracheally intubated ICU patients in need of GFT placement or replacement, who are willing to participate in the study and provide informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Estimated)
Dates: Start 2023-12-18 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Test effectiveness of ultrasound in determining gastric feeding tube position in stomach. | ultrasound control of gastric feeding tube, confirming with X-ray
  To assess the effectiveness of the test we will calculate its sensitivity and specificity. Sensitivity in this case being the proportion of images categorized as having a "mosaic sign present" by the blinded intensivist and indeed representing a gastric GFT localisation (objectivized by CXR). Specificty being the proportion of images categorized as "mosaic sign absent" and representing a non-gastric GFT localisation ( Air insuflation at 20cm GFT insertion and in tracheal canula (TB)). Sensitvity and Specificity will be expressed as a percentage as well as false positive and false negative rates. With this information we will be able to calculate the Likelihood Ratio (LR) for a positive result and for a negative result.
  The analysis will be done using the statistical program SPSS.

SECONDARY OUTCOMES:
Correlating results with basline patient demographic, ventilator settings and post procedure chest x-ray findings. | baseline and post procedure ( gastric feeding tube) chest x-ray
  Correlation of false positive and false negative results with demographic parameters, ventilator settings and chest x-ray findings.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge E Lopez Matta, M.D., Principal Investigator — Leiden University Medical Center
Locations (1):
- Ledien University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlies results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD and supporting information will be available 6 months after publication
Access Criteria: IPD Sharing Access Criteria:
  The anonymized IPD will be shared with qualified researchers affiliated with academic, healthcare institutions, or regulatory authorities, with a focus on diagnostic ultrasound or gastric feeding tube placement. Data will be shared for secondary analyses related to diagnostic methods, ultrasound efficacy, and critical care. Commercial use will require special approval. Requests must include a research proposal, objectives, and ethical approval. Data will be accessed via secure repositories after approval. A committee, including the principal investigator and an independent ethics reviewer, will assess requests based on scientific merit, relevance, and ethical standards. Approved researchers must sign a data-use agreement.

REFERENCES:
- [Background] Gomes GF, Pisani JC, Macedo ED, Campos AC. The nasogastric feeding tube as a risk factor for aspiration and aspiration pneumonia. Curr Opin Clin Nutr Metab Care. 2003 May;6(3):327-33. doi: 10.1097/01.mco.0000068970.34812.8b. PMID 12690267
- [Background] Lo JO, Wu V, Reh D, Nadig S, Wax MK. Diagnosis and management of a misplaced nasogastric tube into the pulmonary pleura. Arch Otolaryngol Head Neck Surg. 2008 May;134(5):547-50. doi: 10.1001/archotol.134.5.547. No abstract available. PMID 18490579
- [Background] Wendell GD, Lenchner GS, Promisloff RA. Pneumothorax complicating small-bore feeding tube placement. Arch Intern Med. 1991 Mar;151(3):599-602. PMID 1848058
- [Background] Wong KW, Chan HH, Wong CP, Chan MY, Chau JCW, Wong TW. Using color flow detection of air insufflation to improve accuracy in verifying nasogastric tube position. Am J Emerg Med. 2017 Feb;35(2):333-336. doi: 10.1016/j.ajem.2016.12.046. Epub 2016 Dec 21. PMID 28038826
- [Background] Vigneau C, Baudel JL, Guidet B, Offenstadt G, Maury E. Sonography as an alternative to radiography for nasogastric feeding tube location. Intensive Care Med. 2005 Nov;31(11):1570-2. doi: 10.1007/s00134-005-2791-1. Epub 2005 Sep 20. PMID 16172849
- [Background] Chenaitia H, Brun PM, Querellou E, Leyral J, Bessereau J, Aime C, Bouaziz R, Georges A, Louis F; WINFOCUS (World Interactive Network Focused On Critical Ultrasound) Group France. Ultrasound to confirm gastric tube placement in prehospital management. Resuscitation. 2012 Apr;83(4):447-51. doi: 10.1016/j.resuscitation.2011.11.035. Epub 2011 Dec 29. PMID 22209831
- [Background] Kim HM, So BH, Jeong WJ, Choi SM, Park KN. The effectiveness of ultrasonography in verifying the placement of a nasogastric tube in patients with low consciousness at an emergency center. Scand J Trauma Resusc Emerg Med. 2012 Jun 12;20:38. doi: 10.1186/1757-7241-20-38. PMID 22691418